CLINICAL TRIAL: NCT03985839
Title: Prospective Multi-Center Post-Market Clinical Follow-up Study to Evaluate Safety and Performance of the MICRORAPTOR REGENESORB, Knotless REGENESORB and Knotless PEEK Suture Anchors (and MINITAPE Sutures) in Shoulder and Hip Arthroscopic Instability Repair
Brief Title: Safety and Performance of MICRORAPTOR™ Suture Anchors in Shoulder and Hip
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018.20.SMD.MRPTKT.PRO
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2023-11

CONDITIONS: Labral Tear, Glenoid; Acetabular Labrum Tear; Bankart Lesions; Anterior Shoulder Instability; SLAP Lesion; Rotator Cuff Tears
Keywords: Microraptor, suture anchor, knotless, Smith and Nephew
MeSH Terms: conditions — Rotator Cuff Injuries; Bankart Lesions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- MICRORAPTOR™ REGENESORB™ Suture Anchor: MICRORAPTOR™ REGENESORB™ Suture Anchor
  Interventions: Device: MICRORAPTOR™ REGENESORB™ Suture Anchor
- MICRORAPTOR™ Knotless REGENESORB™ Suture Anchor: MICRORAPTOR™ Knotless REGENESORB™ Suture Anchor
  Interventions: Device: MICRORAPTOR™ Knotless REGENESORB™ Suture Anchor
- MICRORAPTOR™ Knotless PEEK Suture Anchor: MICRORAPTOR™ Knotless PEEK Suture Anchor
  Interventions: Device: MICRORAPTOR™ Knotless PEEK Suture Anchor

INTERVENTIONS:
Device: MICRORAPTOR™ REGENESORB™ Suture Anchor — Smith & Nephew MICRORAPTOR™ REGENESORB™ Suture Anchor is a fixation device intended to provide secure attachment of soft tissue to bone.
  Groups: MICRORAPTOR™ REGENESORB™ Suture Anchor
Device: MICRORAPTOR™ Knotless REGENESORB™ Suture Anchor — MICRORAPTOR™ Knotless REGENESORB™ Suture Anchor is fixation device, which consists of an anchor on an inserter, and a suture threader. The anchor consists of the following components: a proximal anchor body (REGENESORB™), and a non-absorbable PEEK (Polyether ether ketone) distal anchor tip.
  Groups: MICRORAPTOR™ Knotless REGENESORB™ Suture Anchor
Device: MICRORAPTOR™ Knotless PEEK Suture Anchor — The MICRORAPTOR™ Knotless PEEK Suture Anchor is a class IIb device, which consists of an anchor on an inserter, and a suture threader. The anchor consists of the following components: a proximal anchor body (PEEK), and a non-absorbable PEEK distal anchor tip.
  Groups: MICRORAPTOR™ Knotless PEEK Suture Anchor

SUMMARY:
This is a prospective, multi-center, PMCF study to evaluate the safety and performance of the MICRORAPTOR REGENESORB suture anchors, MICRORAPTOR Knotless REGENESORB suture anchors, and MICRORAPTOR Knotless PEEK suture anchors implanted in 300 subjects needing reattachment of soft tissue to bone.

DETAILED DESCRIPTION:
The purpose of this trial is to assess, by product, safety and performance post-market of the Microraptor Regenesorb, Microraptor Knotless Regenesorb, and Microraptor Knotless PEEK Suture Anchors. Approximately 18 sites (approximately 3 sites for study shoulder group and 3 sites for study hip group, per product) in the United States will participate in the study. This is an open-label study with consecutive enrollment. The study will continue for 24 months from the date that the last subject received the study treatment to the date that the last subject completes the study as planned. The study duration is planned for 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject requires reattachment of soft tissue to bone for the following indications:

  * Shoulder - Capsular stabilization for Bankart repair, Anterior shoulder instability, SLAP lesion repairs, Capsular shift or capsulolabral reconstructions, Biceps tenodesis, Rotator Cuff Repairs (knotless anchors only)
  * Hip - Acetabular labrum repair/reconstruction
* Subject has consented to participate in the study by signing the EC-approved informed consent form.
* Subject is ≥18 years of age at time of surgery.
* Willing and able to make all required study visits.
* Able to follow instructions.

Exclusion Criteria:

* Known hypersensitivity to the implant material. Where material sensitivity is suspected, appropriate tests should be made and sensitivity ruled out prior to implantation.
* Pathological conditions of bone, such as cystic changes or severe osteopenia, which would compromise secure anchor fixation.
* Pathological conditions in the soft tissues to be attached that would impair secure fixation by suture.
* Comminuted bone surface, which would compromise secure anchor fixation.
* Physical conditions which would eliminate, or tend to eliminate, adequate anchor support or retard healing.
* The presence of infection.
* Conditions which would limit the subject's ability or willingness to restrict activities or follow directions during the healing period.
* Currently using tobacco products (cigarette, smokeless tobacco, ecigarettes, vaping etc.).
* Concurrent bilateral surgery.
* Prior MICRORAPTOR REGENESORB, MICRORAPTOR Knotless REGENESORB, or MICRORAPTOR Knotless PEEK implantation.
* Participation in the treatment period of another clinical trial within thirty (30) days of Visit 1, or during the study.
* Women who are pregnant or nursing.
* History of poor compliance with medical treatment.
* Prior ipsilateral surgeries performed on the joint space.
* Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subject requires reattachment of soft tissue to bone for the following indications:
  * Shoulder - Capsular stabilization for Bankart repair, Anterior shoulder instability, SLAP lesion repairs, Capsular shift or capsulolabral reconstructions, Biceps tenodesis, Rotator Cuff Repairs (knotless anchors only)
  * Hip - Acetabular labrum repair/reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Repair failure rate | 6 months
  To assess repair failure rate at 6 months

SECONDARY OUTCOMES:
Repair failure rate | 12 months
  To assess repair failure rate at 12 months
ROWE shoulder score | 6 and 12 months
  ROWE score for shoulder instability is a 3-item instrument completed by the investigator or qualified, delegated study staff. Its questions address the categories of shoulder stability (0 to 50 points), motion (0 to 20 points), and function (0 to 30 points). Scores range from 0 to 100 with a score of 90-100 points indicating an excellent evaluation, 75-89 points indicating a good evaluation, 51-74 points indicating a fair evaluation, and =< 50 points indicating a poor evaluation.
WOSI shoulder score | 6 and 12 months
  Western Ontario Shoulder Instability Index (WOSI) is a subject completed instrument. Its categories include "physical symptoms" (10 items), "sports, recreation, work" (4 items), "pain" (4 items), "lifestyle" (4 items), and "emotion" (3 items), with each category scored from 0 to 100 using a visual analog scale. Overall scores range from 0 to 2100 with a score of 0 indicating better shoulder function and 2100 indicating worse shoulder function.
Constant-Murley Shoulder Scale | 6 and 12 months
  Constant-Murley Shoulder (CMS) scale assesses four aspects related to shoulder pathology; two subjective: pain and activities of daily living (ADL) and two objective: range of motion (ROM) and strength. The subjective components can receive up to 35 points and the objective 65, resulting in a possible maximum total score of 100 points (best function). Pain and ADL are answered by the subject; ROM and strength require a physical evaluation and are answered by the orthopaedic surgeon or the physiotherapist.
HOS-ADL Score | 6 and 12 months
  Hip Outcome Score (HOS) was designed to assess the outcome of treatment intervention for individuals with acetabular tears who may be functioning throughout a wide range of abilities. It is a subject completed measure that consists of an "Activities of Daily Living" (ADL) subscale (17 scored items) and a "Sports" subscale (9 scored items) in which the response options are presented as 5-point Likert scales. Scores for each subscale range from 0% (least function) to 100% (most function).
Modified Harris Hip Score | 6 and 12 months
  Modified Harris Hip Score (mHHS) is a joint specific score that is completed by both the investigator or qualified, delegated study staff and the subject and consists of 10 items covering domains of pain (1 item, 0-44 points), function (7 items, 0-47 points), functional activities, absence of deformity (1 item, 0-4 points), and hip range of motion (2 items, 0-5 points). Scores range from 0 (worse disability) to 100 (less disability).
Adverse Events (AEs) | 12 months
  All adverse events (AEs) and complications occurring from the time of surgical implantation until study termination or study completion including intraoperative adverse events and complications will be collected and reported.
Anchor absorption/replacement by bone (Knotless Regenesorb only) | 6 and 24 months
  MRI performed to determine anchor absorption/replacement by bone at 6 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ozokwere, Study Chair — Smith & Nephew, Inc.
Locations (12):
- United States (12):
  - University of Colorado, Aurora, Colorado
  - Colorado Springs Orthopaedic Group, Colorado Springs, Colorado
  - Holy Cross Orthopedic Institute, Oakland Park, Florida
  - Emory University - Brookhaven, Brookhaven, Georgia
  - Luminis Health Research Institute, Annapolis, Maryland
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oklahoma Sports and Science Orthopedics / The Physician's Group, Oklahoma City, Oklahoma
  - Palmetto/Prisma Health - University of South Carolina Orthopaedics, Columbia, South Carolina
  - Steadman Hawkins Clinic of the Carolinas, Greenville, South Carolina
  - Atlantic Orthopaedic Specialists, Virginia Beach, Virginia
  - Center for Advanced Orthopaedics / Nova Orthopedic & Spine Care, Woodbridge, Virginia
  - Memorial Medical Center, Ashland, Wisconsin

IPD SHARING:
Plan to Share IPD: No